CLINICAL TRIAL: NCT02068443
Title: A Phase 3 Multicenter, Randomized, Double-blind, Parallel-group, Comparative Study When Metformin Hydrochloride 500 mg is Added on to SYR-322 25 mg in Type 2 Diabetic Patients
Brief Title: Comparative Study to Evaluate Efficacy and Safety When Metformin Hydrochloride 500 mg Once Daily is Added on to SYR-322 25 mg in Type 2 Diabetic Patients With Inadequate Glycemic Control Despite Treatment With SYR-322 25 mg in Addition to Diet and Exercise Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-322-MET/CCT-001; JapicCTI-132377 (Other: Japic CTI); U1111-1151-6515 (Registry Identifier: Universal Trial Number)
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Drug therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — alogliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alogliptin Alone (Active Comparator): Alogliptin 25 mg, tablets, orally, once, daily, after breakfast and metformin hydrochloride placebo-matching, tablets, orally, 2 tablets after breakfast and 1 tablet after dinner for 24 weeks.
  Interventions: Drug: Alogliptin; Drug: Metformin hydrochloride Placebo
- Alogliptin + Metformin Hydrochloride QD (Experimental): Alogliptin 25 mg, tablets, orally, once, daily, after breakfast and metformin hydrochloride 500 mg QD (250 mg x 2 tablets, once daily), tablets, orally, once, daily, after breakfast and 1 metformin hydrochloride placebo-matching, tablet, orally, once, daily, after dinner for 24 weeks.
  Interventions: Drug: Alogliptin; Drug: Metformin hydrochloride; Drug: Metformin hydrochloride Placebo
- Alogliptin + Metformin Hydrochloride BID (Active Comparator): Alogliptin 25 mg, tablets, orally, once, daily, after breakfast and metformin hydrochloride 250 mg BID (twice daily), tablets, orally, 1 tablet after breakfast and 1 tablet after dinner and 1 metformin hydrochloride placebo-matching, tablet, orally, once, daily, after breakfast for 24 weeks.
  Interventions: Drug: Alogliptin; Drug: Metformin hydrochloride; Drug: Metformin hydrochloride Placebo

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets
  Other Names: SYR-322; Nesina®
Drug: Metformin hydrochloride — Metformin hydrochloride tablets
  Other Names: Glycoran®
  Arms: Alogliptin + Metformin Hydrochloride BID; Alogliptin + Metformin Hydrochloride QD
Drug: Metformin hydrochloride Placebo — Metformin hydrochloride placebo-matching tablets

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of 24-week treatment with metformin hydrochloride 500 mg once daily added on to alogliptin (SYR-322) 25 mg in type 2 diabetic patients with inadequate glycemic control despite treatment with alogliptin 25 mg in addition to diet and exercise therapy.

DETAILED DESCRIPTION:
The drugs being tested in this study are called alogliptin and metformin hydrochloride. Alogliptin in combination with metformin hydrochloride was being tested to treat people who have Type 2 diabetes mellitus (T2DM) with inadequate glycemic control despite treatment with alogliptin in addition to diet and exercise. This study looked at the efficacy and safety of alogliptin 25 mg once daily (QD) + metformin hydrochloride 500 mg QD compared to alogliptin 25 mg QD + metformin hydrochloride 250 mg twice daily (BID) and alogliptin 25 mg QD administered alone.

The study enrolled 374 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the three treatment groups-which remained undisclosed to the patient and study doctor during the study (unless there was an urgent medical need):

* Alogliptin 25 mg QD + metformin hydrochloride 500 mg QD
* Alogliptin 25 mg QD + metformin hydrochloride 250 mg BID
* Alogliptin 25 mg QD

This multi-center trial was conducted in Japan. The overall time to participate in this study was 36 weeks (12-week screening period and 24-week treatment period). Participants made multiple visits to the clinic including a final visit 24 weeks after the start of study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of type 2 diabetes mellitus.
2. Has a hemoglobin A1c (HbA1c) (National glycohemoglobin standardization program [NGSP]) of ≥6.9% to <10.5% at 8 weeks after the start of the screening period (Week -4).
3. Has an HbA1c (NGSP) difference between 4 weeks after the start of the screening period (Week -8) and 8 weeks after the start of the screening period (Week -4) being within 10.0% (rounded off to the first decimal place) of the value at 4 weeks after the start of the screening period (Week -8).
4. Has been on a certain diet therapy and exercise therapy (if any) during the screening period.
5. Has been receiving alogliptin on a stable dose and regimen (after breakfast, 25 mg/day) during the screening period.
6. In the opinion of investigator or subinvestigator, the participant is considered appropriate to receive a biguanide as an add-on to alogliptin, at the end of the screening period (Week 0).
7. In the opinion of investigator or subinvestigator, the participant is unlikely to require changes in the dose of antihypertensive agents (including discontinuation and suspension) or an additional antihypertensive agent during the study.
8. Is a male and female aged ≥20 years to <75 years. Participants aged ≥65 years to <75 years need to be considered eligible for the enrollment by the investigator or subinvestigator at the end of the screening period (Week 0) taking into consideration the cardiovascular disorders pulmonary function disorders, renal function, hepatic function, etc.
9. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from signing of informed consent throughout the duration of the study.
10. Is treated in outpatient settings during the screening period.
11. In the opinion of the investigator or subinvestigator, the participant is capable of understanding and complying with protocol requirements.
12. Signs and dates a written, informed consent form prior to the initiation of any study procedures.

Exclusion Criteria:

1. Has received other antidiabetic drugs than alogliptin (including insulin preparations and glucagon-like peptidase-1 [GLP-1] analog preparations) during the screening period.
2. Has clinical manifestations of hepatic impairment.
3. Has an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5 × upper limit of normal during the screening period.
4. Has clinical manifestations of renal impairment, including mild impairment.
5. Has a history of lactic acidosis.
6. Has any cardiovascular disease including shock, heart failure, myocardial infarction and pulmonary embolism, any serious pulmonary function disorder, or any other condition predisposing him/her to hypoxemia.
7. Has dehydration or gastrointestinal dysfunction such as diarrhea or vomiting, which may cause dehydrated state.
8. Has malnutrition, starved state, hyposthenia, pituitary gland dysfunction or adrenal insufficiency.
9. Has any serious cardiac disease, any serious cerebrovascular disorder, or any serious pancreatic or hematological disease (eg, the participant requiring inpatient treatment or having been hospitalized for treatment within 24 weeks prior to the start of the screening period).
10. In the opinion of the investigator or subinvestigator, the participant has clinically significant abnormal hematological parameters of hemoglobin, hematocrit, or erythrocytes during the screening period.
11. Has a systolic blood pressure ≥ 180 mmHg or a diastolic blood pressure ≥ 110 mmHg during the screening period.
12. Has a condition requiring insulin for blood glucose control (eg, severe ketosis, diabetic coma or precoma, type 1 diabetes, severe infection, pre- or post-operative condition, or serious trauma).
13. Has any malignancy.
14. Has a history of hypersensitivity or allergies to dipeptidyl-peptidase-4 (DPP-4) inhibitors or biguanides.
15. Is a habitual drinker consuming more than 100 mL of alcohol on average daily.
16. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol dependence.
17. Requires an excluded medication or a prohibited matter during the study.
18. Has received combination therapy of alogliptin benzoate and metformin hydrochloride in a previous clinical study or as a therapeutic agent.
19. Has received any investigational compound within 12 weeks prior to the start of the screening period (Week -12).
20. Is a participant in another clinical study at the time of signing informed consent.
21. If female, the participant is pregnant or lactating; intending to become pregnant between the time of signing informed consent and the end of the study; or intending to donate ova during such period.
22. Is a study site employee, is its immediate family member, is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling), or may consent under duress.
23. Is considered ineligible for the study for any other reason by the investigator or subinvestigator.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (27):
- Japan (27):
  - Nagoya, Aichi-ken
  - Chiba, Chiba
  - Fukuoka, Fukuoka
  - Kitakyushu-shi, Fukuoka
  - Kurume-shi, Fukuoka
  - Aki-gun, Hiroshima
  - Hiroshima, Hiroshima
  - Koga-shi, Ibaraki
  - Mito, Ibaraki
  - Tushiura-shi, Ibaraki
  - Ushiku-shi, Ibaraki
  - Kanazawa, Ishikawa-ken
  - Takamatsu-chi, Kagawa-ken
  - Sendai, Miyagi
  - Ohita-shi, Ohita
  - Okinawa-shi, Okinawa
  - Shimajiri-gun, Okinawa
  - Kashiwara-shi, Osaka
  - Osaka, Osaka
  - Hiki-gun, Saitama
  - Oyama-shi, Tochigi
  - Shimotsuke-shi, Tochigi
  - Koutoh-ku, Tokyo
  - Meguro-ku, Tokyo
  - Sagae-shi, Yamagata
  - Yamagata, Yamagata
  - Yamaguchi, Yamaguchi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 34 investigative sites in Japan from 06 February 2014 (first patient to sign the informed consent form) to 28 February 2015.
Pre-assignment Details: Participants with a diagnosis of Type 2 Diabetes Mellitus were enrolled equally in a 2:2:1 ratio to 1 of 3 treatment groups: alogliptin in combination with 500 mg total dose metformin hydrochloride administered either once a day (QD) or twice a day (BID) and alogliptin alone.
Groups:
- Alogliptin + Metformin Hydrochloride QD: Alogliptin 25 mg, tablets, orally, once, daily, after breakfast and metformin hydrochloride 500 mg QD (250 mg x 2 tablets, once daily), tablets, orally, QD (once daily), after breakfast and 1 metformin hydrochloride placebo-matching, tablet, orally, once, daily, after dinner for 24 weeks.
Period: Overall Study
Arm/Group | Alogliptin Alone | Alogliptin + Metformin Hydrochloride QD | Alogliptin + Metformin Hydrochloride BID
Started | 71 | 152 | 151
Completed | 64 | 146 | 148
Not Completed | 7 | 6 | 3
Not completed — Pretreatment Event/Adverse Event | 0 | 5 | 2
Not completed — Voluntary Withdrawal | 4 | 0 | 1
Not completed — Lack of Efficacy | 2 | 1 | 0
Not completed — Other Reason Not Specified | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alogliptin Alone | Alogliptin + Metformin Hydrochloride QD | Alogliptin + Metformin Hydrochloride BID | Total
Number analyzed (Participants) | 71 | 152 | 151 | 374
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (10.07) | 56.9 (8.79) | 57.6 (9.72) | 57.2 (9.40)
Age, Customized [Number; unit: participants]
  < 65 years | 52 | 119 | 109 | 280
  ≥ 65 years | 19 | 33 | 42 | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 42 | 45 | 106
  Male | 52 | 110 | 106 | 268
Region of Enrollment [Number; unit: participants]
  Japan | 71 | 152 | 151 | 374
Height [Mean (Standard Deviation); unit: cm] | 165.3 (8.89) | 164.6 (8.82) | 164.6 (9.12) | 164.8 (8.94)
Body Weight [Mean (Standard Deviation); unit: kg] | 68.00 (13.702) | 69.48 (13.074) | 69.55 (14.927) | 69.23 (13.943)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.72 (3.764) | 25.61 (4.231) | 25.52 (4.344) | 25.41 (4.196)
Duration of Type 2 Diabetes [Mean (Standard Deviation); unit: years] | 7.73 (4.666) | 7.02 (5.257) | 7.04 (5.380) | 7.16 (5.195)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] | 88.2 (15.99) | 91.0 (16.82) | 87.9 (17.86) | 89.2 (17.11)
Hemoglobin A1c (HbA1c) [National Glycohemoglobin Standardization Program (NGSP)] [Mean (Standard Deviation); unit: percent] | 7.77 (0.780) | 7.82 (0.820) | 7.89 (0.791) | 7.84 (0.800)
Fasting Blood Glucose [Mean (Standard Deviation); unit: mg/dL] | 162.4 (31.03) | 164.7 (31.02) | 165.9 (30.92) | 164.7 (30.92)
Fasting Insulin [Mean (Standard Deviation); unit: μU/mL] | 9.918 (6.8797) | 9.464 (6.7691) | 9.342 (6.0645) | 9.501 (6.4990)
Fasting Glucagon [Mean (Standard Deviation); unit: pg/mL] | 91.7 (30.03) | 86.8 (21.27) | 89.3 (27.98) | 88.8 (25.89)
Homeostasis Model Assessment of Insulin Resistance (HOMA-R) [Mean (Standard Deviation); unit: unitless] | 4.05 (3.238) | 3.87 (2.869) | 3.92 (2.820) | 3.93 (2.916)
Homeostasis Model Assessment Beta Cell Index (HOMA-β) [Mean (Standard Deviation); unit: percent] | 38.64 (29.181) | 36.05 (27.848) | 34.27 (23.638) | 35.82 (26.464)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin A1c (HbA1c) National Glycohemoglobin Standardization Program (NGSP) at the End of Treatment (EOT) Period
Description: The change in the value of HbA1c (NGSP) (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at End of Treatment Period relative to Baseline. A negative change from Baseline indicates improvement. An Analysis of Covariate (ANCOVA) model with change from Baseline as a dependent variable and Baseline and treatment as independent variables was used for main analyses.
Time Frame: Baseline and End of Treatment (EOT) (Up to Week 24)
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Alogliptin Alone | Alogliptin + Metformin Hydrochloride QD | Alogliptin + Metformin Hydrochloride BID
Number analyzed (Participants) | 71 | 152 | 151
percent | 0.16 (0.072) | -0.49 (0.049) | -0.60 (0.049)
Statistical Analysis 1: Comparison: Alogliptin Alone vs Alogliptin + Metformin Hydrochloride QD; Test type: Superiority or Other; LS Mean Difference = -0.65, 95% CI 2-sided [-0.821 to -0.480], Standard Error of Mean 0.087 — Estimated Value was for the difference between Alogliptin + Metformin Hydrochloride QD and Alogliptin alone (Metformin QD - Alogliptin alone)
Statistical Analysis 2: Comparison: Alogliptin + Metformin Hydrochloride QD vs Alogliptin + Metformin Hydrochloride BID; Test type: Non-Inferiority or Equivalence — Non-inferiority of Alogliptin + Metformin Hydrochloride QD to Alogliptin + Metformin Hydrochloride BID; LS Mean Difference = 0.11, 95% CI 2-sided [-0.026 to 0.247], Standard Error of Mean 0.069 — Estimated Value was for the difference between Alogliptin + Metformin Hydrochloride QD and Alogliptin + Metformin Hydrochloride BID (Metformin QD - Metformin BID)

2. Secondary Outcome: Change From Baseline in HbA1c (NGSP)
Description: The change in the value of HbA1c (NGSP) (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Weeks 2, 4, 8, 12, 16, 20, 24, and EOT relative to Baseline. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24 and EOT (Up to Week 24)
Population: FAS, all randomized participants who received at least 1 dose of study drug, with data available for analyses.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Alogliptin Alone | Alogliptin + Metformin Hydrochloride QD | Alogliptin + Metformin Hydrochloride BID
Number analyzed (Participants) | 71 | 152 | 151
percent
  Week 2 (n=71, 152, 151) | 0.01 (0.197) | -0.14 (0.203) | -0.19 (0.212)
  Week 4 (n=70, 150, 150) | 0.01 (0.316) | -0.28 (0.279) | -0.35 (0.298)
  Week 8 (n=68, 149, 149) | -0.01 (0.402) | -0.50 (0.408) | -0.60 (0.454)
  Week 12 (n=67, 148, 148) | -0.02 (0.518) | -0.61 (0.530) | -0.75 (0.565)
  Week 16 (n=66, 148, 147) | 0.01 (0.543) | -0.64 (0.553) | -0.81 (0.602)
  Week 20 (n=65, 146, 148) | 0.11 (0.568) | -0.58 (0.585) | -0.71 (0.626)
  Week 24 (n=64, 146, 148) | 0.17 (0.628) | -0.49 (0.629) | -0.62 (0.659)
  EOT (n=71, 152, 151) | 0.17 (0.616) | -0.49 (0.620) | -0.62 (0.654)

3. Secondary Outcome: HbA1c (NGSP)
Description: The value of HbA1c (NGSP) (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, and EOT.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24 and EOT (Up to Week 24)
Population: FAS, all randomized participants who received at least 1 dose of study drug, with data available for analyses.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Alogliptin Alone | Alogliptin + Metformin Hydrochloride QD | Alogliptin + Metformin Hydrochloride BID
Number analyzed (Participants) | 71 | 152 | 151
percent
  Baseline (n=71, 152, 151) | 7.77 (0.780) | 7.82 (0.820) | 7.89 (0.791)
  Week 2 (n=71, 152, 151) | 7.78 (0.824) | 7.67 (0.796) | 7.70 (0.787)
  Week 4 (n=70, 150, 150) | 7.78 (0.913) | 7.55 (0.773) | 7.54 (0.735)
  Week 8 (n=68, 149, 149) | 7.72 (0.889) | 7.32 (0.725) | 7.28 (0.707)
  Week 12 (n=67, 148, 148) | 7.70 (0.987) | 7.19 (0.721) | 7.13 (0.706)
  Week 16 (n=66, 148, 147) | 7.70 (0.990) | 7.16 (0.725) | 7.08 (0.717)
  Week 20 (n=65, 146, 148) | 7.81 (1.023) | 7.23 (0.749) | 7.18 (0.780)
  Week 24 (n=64, 146, 148) | 7.86 (0.983) | 7.32 (0.798) | 7.27 (0.805)
  EOT (n=71, 152, 151) | 7.95 (1.018) | 7.33 (0.819) | 7.28 (0.804)

4. Secondary Outcome: Percentage of Participants Achieving Target HbA1c (NGSP) Levels at the EOT Period
Description: HbA1c (NGSP) is the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound. The percentage of participants with HbA1c levels of ≥6.0, ≥7.0 and ≥8.0 at the end of Screening (Baseline) with change to target values <6.0, <7.0 and <8.0 respectively at EOT.
Time Frame: Baseline and EOT (Up to Week 24)
Population: FAS included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin Alone | Alogliptin + Metformin Hydrochloride QD | Alogliptin + Metformin Hydrochloride BID
Number analyzed (Participants) | 71 | 152 | 151
percentage of participants
  ≥6.0 at Baseline to <6.0 at EOT (n=71, 152, 151) | 0.0 [lower limit 0.197] | 0.7 [lower limit 0.203] | 1.3 [lower limit 0.212]
  ≥7.0 at Baseline to <7.0 at EOT ( n=63, 137, 140) | 4.8 [lower limit 0.316] | 35.0 [lower limit 0.279] | 34.3 [lower limit 0.298]
  ≥8.0 at Baseline to <8.0 at EOT (n=26, 59, 64) | 23.1 [lower limit 0.402] | 47.5 [lower limit 0.408] | 60.9 [lower limit 0.454]

5. Secondary Outcome: Change From Baseline in Fasting Blood Glucose
Description: The change in the value of the fasting plasma glucose collected at Weeks 2, 4, 8, 12, 16, 20 and 24 relative to Baseline. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24 and EOT (Up to Week 24)
Population: FAS, all randomized participants who received at least 1 dose of study drug, with data available for analyses.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin Alone | Alogliptin + Metformin Hydrochloride QD | Alogliptin + Metformin Hydrochloride BID
Number analyzed (Participants) | 71 | 152 | 151
mg/dL
  Week 2 (n=71, 152, 151) | 0.4 (16.62) | -16.6 (18.99) | -23.7 (20.50)
  Week 4 (n=70, 150, 150) | -0.9 (26.32) | -16.4 (20.79) | -25.2 (20.73)
  Week 8 (n=68, 149, 149) | -2.1 (23.30) | -18.4 (20.90) | -23.4 (24.13)
  Week 12 (n=67, 148, 148) | 1.5 (20.42) | -15.2 (23.83) | -22.9 (24.36)
  Week 16 (n=66, 148, 148) | 0.4 (22.63) | -13.0 (24.70) | -22.6 (25.50)
  Week 20 (n=65, 146, 148) | 6.6 (23.87) | -11.3 (23.34) | -17.6 (25.25)
  Week 24 (n=64, 146, 148) | 8.0 (21.85) | -7.2 (26.53) | -18.2 (25.28)
  EOT (n=71, 152, 151) | 7.4 (26.89) | -7.6 (26.41) | -18.2 (25.41)

6. Secondary Outcome: Fasting Blood Glucose
Description: The value of the fasting plasma glucose collected at Baseline and Weeks 2, 4, 8, 12, 16, 20, 24 and EOT.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24 and EOT (Up to Week 24)
Population: FAS, all randomized participants who received at least 1 dose of study drug, with data available for analyses.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin Alone | Alogliptin + Metformin Hydrochloride QD | Alogliptin + Metformin Hydrochloride BID
Number analyzed (Participants) | 71 | 152 | 151
mg/dL
  Baseline (n=71, 152, 151) | 162.4 (31.03) | 164.7 (31.02) | 165.9 (30.92)
  Week 2 (n=71, 152, 151) | 162.8 (33.42) | 148.1 (26.70) | 142.3 (25.24)
  Week 4 (n=70, 150, 150) | 161.4 (37.17) | 148.7 (27.56) | 140.7 (23.74)
  Week 8 (n=68, 149, 149) | 158.9 (33.15) | 146.5 (25.21) | 142.0 (25.35)
  Week 12 (n=67, 148, 148) | 161.1 (33.43) | 149.2 (30.70) | 142.5 (27.85)
  Week 16 (n=66, 148, 148) | 158.5 (29.71) | 151.4 (32.52) | 142.9 (26.16)
  Week 20 (n=65, 146, 148) | 164.6 (31.64) | 153.2 (30.92) | 147.8 (28.21)
  Week 24 (n=64, 146, 148) | 165.9 (31.19) | 157.4 (33.21) | 147.3 (26.85)
  EOT (n=71, 152, 151) | 169.8 (36.03) | 157.1 (32.82) | 147.7 (27.20)

7. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: 24 Weeks
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin Alone | Alogliptin + Metformin Hydrochloride QD | Alogliptin + Metformin Hydrochloride BID
Number analyzed (Participants) | 71 | 152 | 151
percentage of participants | 57.7 | 50.7 | 52.3

8. Secondary Outcome: Percentage of Participants With TEAEs Categorized Into Investigations System Organ Class (SOC) Related to Chemistry, Hematology or Urinalysis
Description: The percentage of participants with any clinically relevant safety laboratory changes (chemistry, hematology and urinalysis) collected throughout study and recorded as AEs.
Time Frame: 24 Weeks
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin Alone | Alogliptin + Metformin Hydrochloride QD | Alogliptin + Metformin Hydrochloride BID
Number analyzed (Participants) | 71 | 152 | 151
percentage of participants
  Blood Creatine Phosphokinase increased | 0 | 2.0 | 0.7
  Blood Lactic Acid increased | 0 | 1.3 | 0
  Amylase increased | 0 | 0 | 2.0
  Lipase increased | 0 | 0 | 2.0
  Blood Albumin decreased | 0 | 0 | 0.7
  Gamma-glutamyltransferase increased | 0 | 0 | 0.7

9. Secondary Outcome: Percentage of Participants With TEAEs Related to Vital Signs
Description: Vital signs included sitting systolic and diastolic blood pressures (mmHg) (measured after resting for ≥ 5 minutes) and pulse rate (beats per minute [bpm]).
Time Frame: 24 Weeks
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin Alone | Alogliptin + Metformin Hydrochloride QD | Alogliptin + Metformin Hydrochloride BID
Number analyzed (Participants) | 71 | 152 | 151
percentage of participants
  Hypertension | 1.4 | 0 | 0
  Blood Pressure increased | 0 | 0 | 0.7

10. Secondary Outcome: Number of Participants Who Had Clinically Relevant Changes in 12-Lead Electrocardiogram (ECG) Findings
Description: Number of participants who had ECG findings changed from "normal" or "abnormal but not clinically relevant" at Baseline to "abnormal and clinically relevant".
Time Frame: Baseline and Weeks 12 and 24
Population: Safety Analysis Set, all participants who received at least 1 dose of study drug, with ECG values "normal" or "abnormal not clinically significant" at Baseline.
Measure: Number; unit: participants
Arm/Group | Alogliptin Alone | Alogliptin + Metformin Hydrochloride QD | Alogliptin + Metformin Hydrochloride BID
Number analyzed (Participants) | 71 | 151 | 151
participants
  Week 12 | 0 | 0 | 0
  Week 24 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: 24 Weeks
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alogliptin Alone | Alogliptin + Metformin Hydrochloride QD | Alogliptin + Metformin Hydrochloride BID
Serious Adverse Events (participants affected / at risk) | 1/71 | 3/152 | 0/151
Other Adverse Events (participants affected / at risk) | 15/71 | 25/152 | 27/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin Alone (N=71) | Alogliptin + Metformin Hydrochloride QD (N=152) | Alogliptin + Metformin Hydrochloride BID (N=151)
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Splenic injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin Alone (N=71) | Alogliptin + Metformin Hydrochloride QD (N=152) | Alogliptin + Metformin Hydrochloride BID (N=151)
Nasopharyngitis (Infections and infestations) | 8 | 22 | 19
Pharyngitis (Infections and infestations) | 3 | 3 | 9
Hypoaesthesia (Nervous system disorders) | 4 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.